CLINICAL TRIAL: NCT03485521
Title: Interest of High Fidelity Simulation Training Beginning as Part of the Procedure Tracheobronchial Aspiration
Brief Title: Interest of Simulation as Part of the Procedure Tracheobronchial Aspiration
Acronym: SIMREAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/17/0156; 2017-A01609-44 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Tracheobronchial Anomalies
Keywords: High Fidelity Simulation Training; physiotherapy; tracheobronchial aspiration.

STUDY DESIGN:
Intervention Model Description: It is a pilot study, monocentric with randomization of para-medical personnel The randomization list is established by the researcher before the search begins. The strengths of the 3 treatment groups are balanced (15 per group). A document describing the randomization procedure is kept confidential.
Who Masked: Care Provider
Masking Description: The randomization list is established by the researcher before the search begins.
  A document describing the randomization procedure is kept confidential.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practical Work (Active Comparator): 15 students who participate in a practical work lasting two hours about the procedures of the tracheobronchial aspiration
  Interventions: Procedure: The tracheobronchial aspiration
- Stimulation Group (Experimental): Group with competences and reasoning clinic 15 students Simulation with a procedural practice of tracheobronchial suction as part of a simulation sequence after reading the procedures of the tracheobronchial aspiration
  Interventions: Procedure: The tracheobronchial aspiration

INTERVENTIONS:
Procedure: The tracheobronchial aspiration — Reading of the procedures of the tracheobronchial aspiration (legislative framework, rules of hygiene, procedures, undesirable effects) The Practical Group participates in a practical work lasting two hours and the Stimulation Group is in simulation with a procedural practice of tracheobronchial suction as part of a simulation sequence. This group benefits from the methodology of the simulation with a part of briefing, a part simulated session and to finish the debriefing.
  The experiment finished with a real activity on patients with tracheotomy with in this environment the reproduction of the procedure

SUMMARY:
The aim of this study is to compare a control group (Practical Work Group) with a High fidelity Stimulation group about competences and reasoning clinic.

DETAILED DESCRIPTION:
Health simulation is in full development on the national territory (France). The medical profession and nurses use this mode of learning in initial training to improve the students skills The report of Pr Granry allowed an inventory of the simulation in France with as Leitmotiv "never the first time for the patient". It has also put in place priorities for the coming years, one of which is to develop simulation in initial and in-service training. This learning technique is interesting according to several parameters. First,is the safety of care. A novice who has already practiced on a mannequin or in the context of the simulation will be able to better understand the situation of care in the clinical field. The quality of care is also improved by the practice of simulation including communication skills, psychomotor skills, respect for procedures and theoretical knowledge. This more or less faithful reproduction is all the more necessary as the duration of clinical placements is decreasing. Simulation is a way to mitigate this lack is allows a faithful immersion in the care environment. Despite all these positive points, physiotherapy is not yet very affected by the simulation as shown in the literature Gordon's review (2015). Initial training, continuing education has not to this day largely developed this teaching method . Some timid uses have taken place and for the most part in Anglo-Saxon countries with various modes of simulation. In France, certainly linked to the specificity of the profession, its implementation is delicate, even complicated. It remains anecdotal to this day.

ELIGIBILITY:
Inclusion Criteria:

* Learners: All second year students enrolled in initial training of the Institute of kinesitherapy of Toulouse during the year 2017-2018. In total 45 students.
* Patients :All adult patients with tracheotomy, and able to communicate. Patients hospitalized in the University Hospital de Toulouse

Exclusion Criteria:

* Learners: Students absent on the day of the reading of the procedures
* Patients:Adolescent patients, child patients, Patients with a communication deficit, Patients under respirators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-01-13 (Actual); Study Completion 2018-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the acquisition of the skills of a tracheobronchial aspiration procedure | Two hours
  Evaluate the acquisition of the skills of a tracheobronchial aspiration procedure by an audit grid learning according to two different groups (Stimulation group and Practical Work group), on a learner population in initial formation of Institut physiotherapy.

SECONDARY OUTCOMES:
Compare the components of clinical reasoning : self-confrontation and simulation | Two hours
  Compare the components of clinical reasoning in different training typologies : practical work by using simple self-confrontation and simulation The simulation is filmed to watch the action of the learner after with him and bring out the implicit part of the student's clinical reasoning during the performance of the act (self-confrontation).

CONTACTS AND LOCATIONS:
Overall Officials: Didier Alain, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No